CLINICAL TRIAL: NCT04626492
Title: Clinical Study on the Value of Quantitative MRI Imaging in Diffuse Liver Diseases
Brief Title: Quantitative MRI Imaging in Diffuse Liver Diseases
Acronym: QMIDLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, ShaoLin Li, Director of Radiology Department, Fifth Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ZDWY.FSK.005
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Fibrosis and Cirrhosis of Liver
Keywords: Magnetic resonance imaging; Fatty liver; Liver Steatosis; Steatohepatitis; Liver Fibrosis; Hepatic Cirrhosis; Dynamic contrast enhanced magnetic resonance imaging
MeSH Terms: conditions — Fibrosis; Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Such as blood routine,liver function and liver enzyme,renal function, serous markers of liver fibrosis,blood lipid,indicators related to hepatitis virus infection,emergency biochemistry,etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- F0: Normal control group
  Interventions: Diagnostic Test: Quantitative MRI imaging
- F1: Grade 1 of liver fibrosis
  Interventions: Diagnostic Test: Quantitative MRI imaging
- F2: Grade 2 of liver fibrosis
  Interventions: Diagnostic Test: Quantitative MRI imaging
- F3: Grade 3 of liver fibrosis
  Interventions: Diagnostic Test: Quantitative MRI imaging
- F4: Hepatic cirrhosis
  Interventions: Diagnostic Test: Quantitative MRI imaging

INTERVENTIONS:
Diagnostic Test: Quantitative MRI imaging — Dynamic contrast enhanced magnetic resonance imaging,Intravoxel incoherent motion (IVIM) diffusion-weighted magnetic resonance imaging,Iterative decomposition of water and fat with echo asymmetry and least squares estimation quantification sequence

SUMMARY:
As we all know, the early diagnosis and accurate staging of liver fibrosis are very important to reduce the incidence of liver cirrhosis and liver cancer. And the accurate evaluation of hepatic fibrosis is of great significance to the prediction of residual liver function after liver surgery. Therefore, clinicians pay more and more attention to the qualitative and quantitative diagnosis of hepatic fibrosis, liver cirrhosis and hepatic steatosis involved in diffuse liver diseases(such as fatty liver, viral hepatitis, autoimmune hepatitis ). And now, liver biopsy is commonly used as the gold standard for the evaluation of steatohepatitis and fibrosis. However, this test is invasive, has low patient acceptance. So more and more clinicians recommend non-invasive methods to qualitatively and quantitatively evaluate the liver steatosis, fibrosis and cirrhosis in diffuse liver diseases. At present, serum markers, ultrasonic elastography and magnetic resonance imaging have good accuracy in the non-invasive detection and evaluation of liver cirrhosis. However, serum markers are not liver-specific, and a single serum marker is not enough to accurately reflect the degree of liver fibrosis. Furthermore, whether the non-invasive liver fiber diagnostic model is suitable for patients with liver disease in China remains to be further verified. At present, transient elastography has been recommended for the non-invasive staging of hepatic fibrosis by the clinical practice guidelines of the European Association for liver Research and the Asia-Pacific Association for liver Research. But as serum markers, it still has low sensitivity and specificity in the diagnosis of early hepatic fibrosis, and is highly operationally dependent. With the development of MRI technology, some MRI quantitative techniques, such as T1mapping, T2mapping,Intravoxel incoherent motion diffusion-weighted magnetic resonance imaging(IVIM-DWI), dynamic contrast enhanced magnetic resonance imaging(DCE-MRI) can be used to qualitatively and quantitatively diagnosis of liver fat, hepatic fibrosis and cirrhosis. And iterative decomposition of water and fat with echo asymmetry and least squares estimation quantification sequence(IDEALIQ) usually used to evaluate liver fat. The existing research results showed that MRI quantitative techniques has a high value in quantitative diagnosis of advanced hepatic fibrosis and cirrhosis. But it still has some limitations in quantitative diagnosis of early liver fibrosis. And what's more,some of the research results still can not reach a consensus. Therefore, based on the multi-parameter potential of MRI and the characteristics of metabolic evaluation. This study will adjust some of the parameters of MRI quantitative techniques, and through large sample datas, combined with a variety of quantitative techniques to explore the application value of MRI quantitative techniques in the quantitative diagnosis of liver diffuse lesions, especially in the early stage of liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

Selection criteria for case group (F1-F4) (meet all the following 1-5 criteria can be selected or only meet the 6 criteria)

1. Fatty liver, liver fibrosis or cirrhosis confirmed by clinical, biochemical, imaging examination and liver biopsy;
2. no secondary portal hypertension and increase alpha feto protein(AFP);
3. no thrombus or plaque in the portal vein and abdominal aorta;
4. no history of psychotropic drug addiction;
5. MRI examination three days before liver puncture or liver transplantation;
6. isolated liver of patients undergoing liver transplantation.

The selection criteria of the normal control group (F0) (meet all the following 1-4 criteria can be selected or only meet the 5 criteria):

1. no known acute or chronic liver disease (serologically negative);
2. no history of alcoholism, and normal liver function tests;
3. no signs of chronic liver disease in CT or MRI;
4. no CT or MRI manifestations of focal or diffuse liver disease in the liver;
5. abandoned donor liver

Exclusion Criteria:

1. contraindications for MRI or patients' inability to cooperate with MRI;
2. allergy to contrast media and poor image quality can not meet the needs of clinical diagnosis;
3. less than 18 years of age, poor quality of liver biopsy;
4. renal insufficiency (eGFP < 60ml/min/1.73mm2);
5. with severe heart, brain, lung and blood system diseases.
6. liver complicated with fulminant liver failure and gastrointestinal bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All suspected patients with diffuse liver diseases meet the inclusion criteria will include in this study. And patients who meet the criteria of the normal control group will include in this study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative MRI imaging diagnose diffuse hepatic lesions | 2 years
  Quantitative MRI imaging(such as dynamic contrast enhanced magnetic, intravoxel incoherent motion (IVIM) diffusion-weighted magnetic resonance imaging resonance imaging, Intravoxel incoherent motion (IVIM) diffusion-weighted magnetic resonance imaging, Iterative decomposition of water and fat with echo asymmetry and least squares estimation quantification sequence) used to quantitative diagnosis of fatty liver hepatitis, liver fibrosis, cirrhosis, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shaolin Li, Director, Principal Investigator — Radiology Department，the Fifth Affiliated Hospital of Sun Yat-sen University
Locations (1):
- 52 Meihua East Road, New Xiangzhou, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan JG, Kim SU, Wong VW. New trends on obesity and NAFLD in Asia. J Hepatol. 2017 Oct;67(4):862-873. doi: 10.1016/j.jhep.2017.06.003. Epub 2017 Jun 19. PMID 28642059
- [Background] Sheka AC, Adeyi O, Thompson J, Hameed B, Crawford PA, Ikramuddin S. Nonalcoholic Steatohepatitis: A Review. JAMA. 2020 Mar 24;323(12):1175-1183. doi: 10.1001/jama.2020.2298. PMID 32207804
- [Background] Younossi ZM, Stepanova M, Afendy M, Fang Y, Younossi Y, Mir H, Srishord M. Changes in the prevalence of the most common causes of chronic liver diseases in the United States from 1988 to 2008. Clin Gastroenterol Hepatol. 2011 Jun;9(6):524-530.e1; quiz e60. doi: 10.1016/j.cgh.2011.03.020. Epub 2011 Mar 25. PMID 21440669
- [Background] Poynard T, Lenaour G, Vaillant JC, Capron F, Munteanu M, Eyraud D, Ngo Y, M'Kada H, Ratziu V, Hannoun L, Charlotte F. Liver biopsy analysis has a low level of performance for diagnosis of intermediate stages of fibrosis. Clin Gastroenterol Hepatol. 2012 Jun;10(6):657-63.e7. doi: 10.1016/j.cgh.2012.01.023. Epub 2012 Feb 14. PMID 22343514
- [Background] Dong XQ, Wu Z, Zhao H, Wang GQ; China HepB-Related Fibrosis Assessment Research Group. Evaluation and comparison of thirty noninvasive models for diagnosing liver fibrosis in chinese hepatitis B patients. J Viral Hepat. 2019 Feb;26(2):297-307. doi: 10.1111/jvh.13031. Epub 2018 Nov 28. PMID 30380170
- [Background] Wai CT, Greenson JK, Fontana RJ, Kalbfleisch JD, Marrero JA, Conjeevaram HS, Lok AS. A simple noninvasive index can predict both significant fibrosis and cirrhosis in patients with chronic hepatitis C. Hepatology. 2003 Aug;38(2):518-26. doi: 10.1053/jhep.2003.50346. PMID 12883497
- [Background] Thiele M, Detlefsen S, Sevelsted Moller L, Madsen BS, Fuglsang Hansen J, Fialla AD, Trebicka J, Krag A. Transient and 2-Dimensional Shear-Wave Elastography Provide Comparable Assessment of Alcoholic Liver Fibrosis and Cirrhosis. Gastroenterology. 2016 Jan;150(1):123-33. doi: 10.1053/j.gastro.2015.09.040. Epub 2015 Oct 3. PMID 26435270
- [Background] Wu S, Yang Z, Zhou J, Zeng N, He Z, Zhan S, Jia J, You H. Systematic review: diagnostic accuracy of non-invasive tests for staging liver fibrosis in autoimmune hepatitis. Hepatol Int. 2019 Jan;13(1):91-101. doi: 10.1007/s12072-018-9907-5. Epub 2018 Nov 15. PMID 30443702
- [Background] Zhang YN, Fowler KJ, Hamilton G, Cui JY, Sy EZ, Balanay M, Hooker JC, Szeverenyi N, Sirlin CB. Liver fat imaging-a clinical overview of ultrasound, CT, and MR imaging. Br J Radiol. 2018 Sep;91(1089):20170959. doi: 10.1259/bjr.20170959. Epub 2018 Jun 6. PMID 29722568
- [Background] Singh S, Venkatesh SK, Wang Z, Miller FH, Motosugi U, Low RN, Hassanein T, Asbach P, Godfrey EM, Yin M, Chen J, Keaveny AP, Bridges M, Bohte A, Murad MH, Lomas DJ, Talwalkar JA, Ehman RL. Diagnostic performance of magnetic resonance elastography in staging liver fibrosis: a systematic review and meta-analysis of individual participant data. Clin Gastroenterol Hepatol. 2015 Mar;13(3):440-451.e6. doi: 10.1016/j.cgh.2014.09.046. Epub 2014 Nov 20. PMID 25305349
- [Background] Li Z, Sun J, Chen L, Huang N, Hu P, Hu X, Han G, Zhou Y, Bai W, Niu T, Yang X. Assessment of liver fibrosis using pharmacokinetic parameters of dynamic contrast-enhanced magnetic resonance imaging. J Magn Reson Imaging. 2016 Jul;44(1):98-104. doi: 10.1002/jmri.25132. Epub 2015 Dec 28. PMID 26707910
- [Background] Wu CH, Ho MC, Jeng YM, Liang PC, Hu RH, Lai HS, Shih TT. Assessing hepatic fibrosis: comparing the intravoxel incoherent motion in MRI with acoustic radiation force impulse imaging in US. Eur Radiol. 2015 Dec;25(12):3552-9. doi: 10.1007/s00330-015-3774-4. Epub 2015 May 20. PMID 25991478
- [Background] Li J, Liu H, Zhang C, Yang S, Wang Y, Chen W, Li X, Wang D. Native T1 mapping compared to ultrasound elastography for staging and monitoring liver fibrosis: an animal study of repeatability, reproducibility, and accuracy. Eur Radiol. 2020 Jan;30(1):337-345. doi: 10.1007/s00330-019-06335-0. Epub 2019 Jul 23. PMID 31338650
- [Background] Hoffman DH, Ayoola A, Nickel D, Han F, Chandarana H, Shanbhogue KP. T1 mapping, T2 mapping and MR elastography of the liver for detection and staging of liver fibrosis. Abdom Radiol (NY). 2020 Mar;45(3):692-700. doi: 10.1007/s00261-019-02382-9. PMID 31875241
- [Background] Loomba R, Neuschwander-Tetri BA, Sanyal A, Chalasani N, Diehl AM, Terrault N, Kowdley K, Dasarathy S, Kleiner D, Behling C, Lavine J, Van Natta M, Middleton M, Tonascia J, Sirlin C; NASH Clinical Research Network. Multicenter Validation of Association Between Decline in MRI-PDFF and Histologic Response in NASH. Hepatology. 2020 Oct;72(4):1219-1229. doi: 10.1002/hep.31121. Epub 2020 Oct 9. PMID 31965579